CLINICAL TRIAL: NCT01565200
Title: Phase II Prospective Imaging Study Evaluating the Utility of Pre-treatment zr89 Labelled Trastuzumab PET/CT and an Early FDG-PET/CT Response to Identify Patients With Advanced HER2+ BC Unlikely to Benefit From a Novel antiHER2 Therapy: TDM1
Brief Title: HER2 Imaging Study to Identify HER2 Positive Metastatic Breast Cancer Patient Unlikely to Benefit From T-DM1
Acronym: ZEPHIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJBMNTDM1; 2011-005437-39 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-28 (Estimated); Last update posted 2025-03-31 (Actual); Status verified 2022-11

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: HER2; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; zirconium-89-trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T-DM1 (Other): After an imaging phase, the patient will receive T-DM1 iv every 3 weeks until progression or toxicity
  Interventions: Drug: T-DM1; Procedure: 89Zr-trastuzumab

INTERVENTIONS:
Drug: T-DM1 — 3.6 mg/kg iv every 3 weeks
  Other Names: Trastuzumab-DM1
Procedure: 89Zr-trastuzumab — Injection of 89Zr-trastuzumab for HER2 imaging
  Other Names: Zirconium 89 labelled trastuzumab

SUMMARY:
T-DM1 , which is a highly innovative but also expensive antiHER2 agent consisting in the coupling of the humanised monoclonal antibody trastuzumab with a cytotoxic agent (maytansine derivate) has shown an encouraging antitumor activity evaluated by Recist criteria (35% objective response rate, 44% stable disease, 18% progressive disease) in patients with advanced HER2 positive Breast Cancer pretreated with several cytotoxic drugs, trastuzumab and lapatinib.

Rationale I :For TDM1 to be active, the presence of an intact HER2 receptor is "key" since the internalization of the cytotoxic moiety depends on the binding of trastuzumab to the external domain of HER2.

The zirconium 89 labelled trastuzumab PET/CT (or HER2 immunoPET/CT) is a non invasive test which shows promise in measuring HER2 expression (extracellular domain) for the entire disease burden and which could identify non responding patients prior to TDM1 administration.

Rationale II: As for many such agents, it is desirable to identify early on (here with the use of FDG-PET/CT) which patients are unlikely to benefit from the therapy

DETAILED DESCRIPTION:
The main objective of the trial is to prospectively evaluate the ability of a zirconium 89 labelled trastuzumab PET, to predict, before initiation of the treatment, treatment failure to a new targeted drug: T-DM1.

At the same time, the early FDG-PET/CT, performed after 1 course of T-DM1, will also evaluated for its ability to predict non response to TDM1.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have histologically confirmed HER2 positive invasive carcinoma of the breast in the reference laboratory of the participating center. HER2 positive criteria to be applied are those used in the participating countries:

   * Belgium: FISH amplification ratio ≥ 2 in the reference laboratory of the participating center
   * The Netherlands: IHC 3+ or FISH ratio ≥ 2 in the reference laboratory of the participating center
2. The patient must have documented progressive disease and present with at least 2 non-bone "target" metastatic lesions, unequivocally of neoplastic origin with

   * a transaxial diameter greater than 2 cm on the screening diagnostic CT/MRI for all non-bone lesions except lymphnodes
   * a short axis greater than 1,5 cm for lymphnodes on the screening diagnostic CT/MRI These two lesions should not be confluent with adjacent lesions and not have been irradiated previously.
3. A concurrent biopsy of a metastatic site is mandatory (with two formalin fixed paraffin embedded (FFPE) core sample and two snap frozen tumor sample) after progression has been documented and before inclusion and the patient agrees with the procedure.
4. Primary tumor blocks (or 11 unstained slides) available for confirmatory central laboratory HER2 testing in Institut Jules Bordet. If available, a snap frozen sample of the primary tumor will also be centralized in Institut Jules Bordet.
5. Age ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1
7. No significant cardiac history and current LVEF ≥ 50%
8. Adequate organ function, evidenced by the following laboratory results:

   * Absolute neutrophil count > 1,500 cells/mm3
   * Platelet count > 100,000 cells/mm3
   * Hemoglobin > 9 g/dL
   * AST(SGOT) and ALT (SGPT) < 2.5 x ULN
   * Total Bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert's syndrome. Patients with known Gilbert's Syndrome should have direct bilirubin within normal limits.
   * Serum alkaline phosphatase ≤ 2.5 x ULN. Patients with bone metastases: alkaline phosphatase ≤ 5 x ULN
   * Serum creatinine < 2.0 mg/dL or 177 μmol/L
   * International normalized ratio (INR) and activated partial thromboplastin time or partial thromboplastin time (aPTT or PTT) < 1.5 x ULN (unless on therapeutic anti-coagulation except vitamin K antagonists which are prohibited in this study)
9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
10. For women of childbearing potential a serum pregnancy test will be done (and it must be negative) and an agreement to use a highly-effective form of contraception during all the study and at least the following 7 months will be obtained.
11. Signed written informed consent obtained prior to any study specific procedure.
12. Completion of all necessary baseline surgical, laboratory and imaging investigations prior to patient inclusion.

Exclusion Criteria:

1. Patients with bone only metastases are not eligible.
2. Diffuse liver (≥50%) involvement on imaging.
3. Patients with brain metastasis as the sole site of metastatic disease and/or are symptomatic or require therapy to control symptoms NB: Brain metastasis are allowed provided they are asymptomatic and/or controlled by previous radiotherapy. In case of recent prior brain radiotherapy, there must be evidence on MRI imaging of brain metastatic control for at least 6 weeks since the end of radiotherapy. Moreover, the patient should be at the end of corticosteroid therapy and be clinically asymptomatic.
4. Current uncontrolled hypertension despite medication intake (systolic > 150 mmHg and/or diastolic > 100 mmHg)
5. Current unstable angina
6. History of symptomatic CHF of any New York Heart Association (NYHA) criteria or ventricular arrhythmia that requires treatment
7. History of myocardial infarction within the last 6 months
8. History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
9. Current dyspnea at rest due to complications of advanced malignancy, or other diseases that require continuous oxygen therapy
10. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures)
11. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those previously mentioned
12. Pregnant or lactating women
13. Concurrent, serious, uncontrolled infections or current known infection with HIV, active hepatitis B and/or hepatitis C.
14. Known prior severe hypersensitivity to trastuzumab
15. Patient who received lapatinib within the 15 days prior to 89Zr-Trastuzumab injection
16. Patient under a prohibited concomitant therapy, including vitamine K antagonist
17. Patients with a peripheral neuropathy Grade 3 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
negative predictive value of the 89Zr-trastuzumab PET/CT | 2 years
  The primary objective is to show that pre-treatment 89Zr-trastuzumab PET/CT is able to select lesions not responding morphologically from treatment with T-DM1 (applying RECIST 1.0 criteria).

SECONDARY OUTCOMES:
negative predictive value of the early FDG PET/CT | 2 years
  The first secondary objective is to show that early FDG PET/CT (performed after one cycle of T-DM1 just before the second cycle) is able to select lesions not responding from treatment with T-DM1 according to metabolic and morphological response criteria post 3 cycles of T-DM1.
negative predictive value of the 89Zr-trastuzumab PET/CT | 2 years
  The second secondary objective is to show that 89Zr-trastuzumab PET/CT is able to select lesions not responding from treatment with T-DM1 according to metabolic response criteria post 3 cycles of T-DM1.
negative predictive value of the combined 89Zr-trastuzumab PET/CT and early PET/CT | 2 years
  The third secondary objective is to show that a lesion with no/faint uptake on 89Zr-trastuzumab PET/CT and not responding metabolically on the early FDG-PET/CT will not respond according to metabolic and morphological criteria after 3 cycles of T-DM1.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flamen, MD/PhD, Study Chair — Jules Bordet Institute
Locations (5):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Antwerp, Edegem
  - Institut Jules Bordet, Brussels
- Netherlands (3):
  - Vrije Universiteit Amsterdam (VUMC), Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud University Medical Centre Nijmegen (UMCN), Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gebhart G, Lamberts LE, Wimana Z, Garcia C, Emonts P, Ameye L, Stroobants S, Huizing M, Aftimos P, Tol J, Oyen WJ, Vugts DJ, Hoekstra OS, Schroder CP, Menke-van der Houven van Oordt CW, Guiot T, Brouwers AH, Awada A, de Vries EG, Flamen P. Molecular imaging as a tool to investigate heterogeneity of advanced HER2-positive breast cancer and to predict patient outcome under trastuzumab emtansine (T-DM1): the ZEPHIR trial. Ann Oncol. 2016 Apr;27(4):619-24. doi: 10.1093/annonc/mdv577. Epub 2015 Nov 23. PMID 26598545